CLINICAL TRIAL: NCT06067100
Title: Physiological Response to U-LABA/ICS With Emphasis on Exercise Performance, Indacaterol
Brief Title: U-LABA/ICS Effects on Exercise Performance, Indacaterol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: INDAC
Record Dates: First submitted 2023-09-20; First posted 2023-10-04 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Exercise Performance
MeSH Terms: interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Indacaterol + mometasonefluroate (Experimental)
  Interventions: Drug: Indacaterol and Mometasonefluroate (low dose); Drug: Indacaterol and Mometasonefluroate (high dose)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol and Mometasonefluroate (low dose) — Participants are administered 125 µg indacaterol + mometasonefluroate
  Arms: Indacaterol + mometasonefluroate
Drug: Placebo — Participants are administered placebo
  Arms: Placebo
Drug: Indacaterol and Mometasonefluroate (high dose) — Participants are administered 500 µg indacaterol + mometasonefluroate
  Arms: Indacaterol + mometasonefluroate

SUMMARY:
The purpose of the project is to investigate exercise performance in humans following bronchodilation induced by acute inhalation of beta2-agonist indacaterol + mometasonefuroate

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39
* Physically active > 5 h weekly
* Maximal oxygen consumption classified as high or very high

Exclusion Criteria:

* Diagnosed with severe asthma and been in treatment with long-acting beta2-agonist/corticosteroid
* ECG abnormality
* ACQ score > 1.5
* Severe bronchial hyperreactivity as determined by mannitol test
* FEV1/FVC ratio < 0.7 determined with spirometry
* Chronic illness determined to be a potential risk for participant during study
* In chronic treatment with medication that may interfere with study results
* Pregnancy
* Smoker
* Blood donation during the past 3 months

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Power output during sprint testing | Through study completion, an average of 3 weeks
  Power output measured in Watts during a sprint on a bike ergometer

SECONDARY OUTCOMES:
Power output during time trial | Through study completion, an average of 3 weeks
  Mean power output measured in Watts during a time trial on a bike ergometer
Forced Expiratory Volume in 1 second (FEV1) | Through study completion, an average of 3 weeks
  FEV1 measured by spirometry
Quadriceps strength | Through study completion, an average of 3 weeks
  Maximal torque (Nm) achieved during isometric contraction
Respiratory muscle function | Through study completion, an average of 3 weeks
  Mouth inspiratory and expiratory pressures (MD Diagnostics, RP-check, handheld respiratory pressure meter)

CONTACTS AND LOCATIONS:
Overall Officials: Morten Hostrup, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided